CLINICAL TRIAL: NCT04488107
Title: A Multicenter, Open, Single Arm Dose-escalation and Dose-expansion Study: to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of FCN-437c Alone or in Combination With Letrozole in ER+/ HER2- Advanced Breast Cancer
Brief Title: Safety, Tolerability, Pharmacokinetics and Antitumor Activity of FCN-437c
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Collaborators: Fudan University (Other); Zhejiang Cancer Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AH150201
Record Dates: First submitted 2020-07-13; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasms
Keywords: ER-Positive; HER2-Negative; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — FCN-437c; Letrozole

STUDY DESIGN:
Intervention Model Description: This study plans to start dose escalating from 50 mg, followed by 100, 200, 300, 450, and 600 mg as tentatively designated escalating dose groups. After the initial dose group, it is allowed to adjust the subsequent dose level according to the test data, but it will not exceed 100% dose increment. After the completion of DLT observation in each group, the next dose group and the number of cases were determined according to the safety, efficacy and PK data of the dose group. The traditional "3+3" method was used in the design of dose escalating stage, and the improved Fibonacci series was used for the dose increasing stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation cohort of FCN-437c (Experimental): * This study plans to start escalating from 50 mg QD, through 100 mg, 200 mg, 300 mg, 450 mg, to 600 mg.
  * Participants will receive FCN-437c in sequential 28-day cycles which are made up of monotherapy QD for 21 days followed by a 7 day rest period.
  * Participants must be histologically or cytologically diagnosed with ER+/ HER2- advanced breast cancer.
  Interventions: Drug: FCN-437c
- Dose expansion cohort of FCN-437c + letrozole (Experimental): * The dose expansion stage will be initiated after escalating to MTD.
  * Six patients will be treated with FCN-437c combined with letrozole.
  * DLT assessment and PK blood collection will be completed in the first 28-day cycle.
  * If DLT does not occur in the first three patients, 15 additional patients were enrolled to complete the expansion study of MTD group.
  * If one DLT occurs in the first three patients, three additional patients will be enrolled onal patients were enrolled and completed the MTD group.
  * Patients will be evaluated every 8 weeks until disease progression, intolerable toxicity, death, investigator's decision or patient's voluntary withdrawal from the study.
  Interventions: Drug: FCN-437c; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: FCN-437c — - FCN-437c is a selective and potent CDK4/6 dual inhibitor, with broad antitumor activity in preclinical pharmacology models, favorable physical and pharmacokinetic (PK) properties, and acceptable toxicity profile in nonclinical studies.
  Other Names: Dose-escalation and expansion
Drug: Letrozole 2.5mg — * Letrozole is the latest generation of aromatase inhibitor. Letrozole lowers estrogen levels in postmenopausal women, which may slow the growth of certain types of breast tumors that need estrogen to grow in the body.
  * Letrozole is used to treat breast cancer in postmenopausal women. It is often given to women who have been taking tamoxifen (Nolvadex, Soltamox) for 5 years.
  Other Names: Dose-escalation
  Arms: Dose expansion cohort of FCN-437c + letrozole

SUMMARY:
This is a multicenter, open, single arm dose escalation and dose expansion clinical study to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of FCN-437c alone or in combination with letrozole in women with ER +/ HER2 - advanced breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, open, single arm clinical study to evaluate the safety, tolerability, and antitumor activity of FCN-437c in combination with letrozole in postmenopausal women with ER + / HER2 - advanced breast cancer, and to evaluate the PK characteristics of FCN-437c monotherapy and combined therapy.

The single drug administration period (7 days) . The continuous administration period made up of 21 days of continuous administration, followed by 7 days of withdrawal, which made up of 28 days as a treatment cycle. The evaluation was conducted every 8 weeks until one of the following happened, disease progression, intolerable toxicity, death, the researcher's decision or the patients' voluntary withdrawal from the study. The follow-up visit was conducted 30 days after the last administration. The telephone follow-up was conducted once every 3 months until the end of the study to record the survival period.

In the expansion period, FCN-437c was continuous administration per day for 21 days, followed by 7 days of withdrawal, making a treatment cycle of 28 days during which letrozole was continuously administrated 2.5 mg QD. Evaluation was conducted every 8 weeks until one of the following occurred, disease progression, intolerable toxicity, death, decision of the researcher or patients' voluntary withdrawal of the study. Follow up visit was conducted 30 days after the last administration, followed by the survival period telephone follow-up every 3 months until the end of the study.

End of of the study was defined as the last patient in the dose expansion stage took the treatment for more than one year, or terminated the treatment (depending on which occurred earlier.

At the end of the study, patients with no disease progression were determined to continue taking FCN-437c according to the clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>= 18 years old) patients diagnosed as ER +/ HER2 - advanced breast cancer, without standard treatment or unable to receive standard treatment;
* The eastern cooperative oncology group (ECOG) score is 0 or 1;
* According to RECIST version 1.1, there was at least one measurable lesion or only bone metastasis;
* The expected survival period is at least 12 weeks;
* Patients have sufficient bone marrow and organ function;
* Patients is willing and able to follow the planned visit, treatment plan, laboratory examination and other test procedures;
* Patients fully understand the study and are willing to sign the informed consent form (ICF);
* The inclusion criteria specific for the dose expansion stage are as follows.
* The postmenopausal patients (>= 18 years old) diagnosed as ER +/ HER2 - breast cancer have evidence of local recurrence or metastasis, and are not suitable for surgical resection or radiotherapy for the purpose of cure;
* There was neither history of systematic treatment nor clinical indication for chemotherapy for patients in the dose expansion stage;
* The patients in the dose expansion stage should neither have received neoadjuvant or adjuvant endocrine therapy previously, nor have progression free survival during or after the neoadjuvant or adjuvant endocrine therapy was shorter than 12 months.

Exclusion Criteria:

* HER2 + breast cancer, either defined as by fluorescence hybridization (FISH) or detected by standard immunohistochemistry (IHC);
* History of previous CDK4 / 6 inhibitors treatment;
* Received anti-tumor chemotherapy, major surgery, radiotherapy, biological drug therapy or other research drug treatment within 28 days before enrollment;
* The toxicity of previous anti-tumor therapy has not recovered (>= grade 2 according to NCI CTCAE version 5.0), except for hair loss; the neurotoxicity of patients who have received chemotherapy before should be restored to grade 2 or below based on NCI CTCAE version 5.0;
* The patient used CYP3A strong inhibitor or CYP3A inducer 14 days before the first dose administration;
* Cardiac dysfunction or disease are consistent with one of the following conditions such as arrhythmia with clinical significance, any risk factors increasing risk of QTc interval prolongation, or congestive heart failure (CHF) with grade ≥ 3 according to NYHA ;
* Dysphagia, active digestive system disease, major gastrointestinal surgery, malabsorption syndrome, or other conditions that may impair the absorption of FCN-437c;
* Known allergy to letrozole, FNC-437c or any other excipients;
* Uncontrolled central system metastasis;
* Active infection, including HBV, HCV, HIV, et al;
* Any other disease or condition of clinical significance (e.g., uncontrolled diabetes, active or uncontrollable infection) that the researchers believe may affect protocol compliance or affect patients' signing of ICF;
* The exclusion criteria specific for the dose expansion stage was as follows.
* Postmenopausal women with advanced breast cancer who have received neoadjuvant / adjuvant endocrine therapy and progressed less than 12 months after treatment;
* Patients with advanced breast cancer who had received systemic anti-tumor therapy including endocrine and chemotherapy (patients with ER + and HER2 - who had received aromatase inhibitors for no more than 14 days were allowed to be enrolled) ;
* Other exclusion criteria are the same as those of the dose escalation stage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer,
Enrollment: 78 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
DLT within 7 days of FCN-437c monotherapy | 7 days
  The incidence of DLT occurred within 7 days of FCN-437c monotherapy
DLT within 28 days of FCN-437c monotherapy | 28 days
  The incidence of DLT occurred within 28 days of FCN-437c monotherapy
DLT within 28 days of FCN-437c combined therapy | 28 days
  The incidence of DLT occurred within 28 days of the letrozole-combined treatment.
Adverse events until the last followup | through study completion, assessed up to 24 months
  The types and frequencies of adverse events (AEs) evaluated according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0.
Serious and significant adverse events | through study completion, assessed up to 24 months
  Serious adverse events (SAE) and toxic reactions leading to permanent drug withdrawal occurred during the treatment.
Incidence of Deaths | through study completion, assessed up to 24 months
  The frequency and causes of deaths during the treatment.
Incidence of abnormal laboratory results | through study completion, assessed up to 24 months
  Abnormal laboratory results of safety concerns such as ALT, AST, Cr and BUN, et al according to NCI-CTCAE 5.0 classification.
Changes of ECGs from baselines | through study completion, assessed up to 24 months
  Changes of ECGs from baselines, such as QT interval。

SECONDARY OUTCOMES:
Anti-tumor efficacy of monotherapy | through study completion, assessed up to 24 months
  Objective response rate (ORR) of FCN-437c monotherapy.
Anti-tumor efficacy of combined treatment | through study completion, assessed up to 24 months
  Objective response rate (ORR) of FCN-437c and letrozole-combined treatment.
FPS | through study completion, assessed up to 24 months
  Progression free survival (PFS) during the treatment.
OS | through study completion, assessed up to 24 months
  overall survival (OS) during the treatment.
survival rate | through study completion, assessed up to 24 months
  1-year OS rate during the 1st year of treatment.
DOR | through study completion, assessed up to 24 months
  duration of response (DOR) during the treatment.
CBR | through study completion, assessed up to 24 months
  clinical benefit response (CBR) during the treatment.
Cmax of FCN-437c in monotherapy | through study completion, assessed up to 24 months
  Maximal plasma concentration of FCN-437c in monotherapy.
AUC of FCN-437c in monotherapy | through study completion, assessed up to 24 months
  Entire exposure of FCN-437c in monotherapy.
Cmax of FCN-437c in combined treatment | through study completion, assessed up to 24 months
  Maximal plasma concentration of FCN-437c combined with letrozole.
AUC of FCN-437c in combined treatment | through study completion, assessed up to 24 months
  Entire exposure of FCN-437c combined with letrozole.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Background] Curigliano G, Gomez Pardo P, Meric-Bernstam F, Conte P, Lolkema MP, Beck JT, Bardia A, Martinez Garcia M, Penault-Llorca F, Dhuria S, Tang Z, Solovieff N, Miller M, Di Tomaso E, Hurvitz SA. Ribociclib plus letrozole in early breast cancer: A presurgical, window-of-opportunity study. Breast. 2016 Aug;28:191-8. doi: 10.1016/j.breast.2016.06.008. Epub 2016 Jun 20. PMID 27336726
- [Background] Infante JR, Cassier PA, Gerecitano JF, Witteveen PO, Chugh R, Ribrag V, Chakraborty A, Matano A, Dobson JR, Crystal AS, Parasuraman S, Shapiro GI. A Phase I Study of the Cyclin-Dependent Kinase 4/6 Inhibitor Ribociclib (LEE011) in Patients with Advanced Solid Tumors and Lymphomas. Clin Cancer Res. 2016 Dec 1;22(23):5696-5705. doi: 10.1158/1078-0432.CCR-16-1248. Epub 2016 Aug 19. PMID 27542767
- [Background] Tamura K, Mukai H, Naito Y, Yonemori K, Kodaira M, Tanabe Y, Yamamoto N, Osera S, Sasaki M, Mori Y, Hashigaki S, Nagasawa T, Umeyama Y, Yoshino T. Phase I study of palbociclib, a cyclin-dependent kinase 4/6 inhibitor, in Japanese patients. Cancer Sci. 2016 Jun;107(6):755-63. doi: 10.1111/cas.12932. Epub 2016 May 11. PMID 26991823
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Elsasser A, Regnstrom J, Vetter T, Koenig F, Hemmings RJ, Greco M, Papaluca-Amati M, Posch M. Adaptive clinical trial designs for European marketing authorization: a survey of scientific advice letters from the European Medicines Agency. Trials. 2014 Oct 2;15:383. doi: 10.1186/1745-6215-15-383. PMID 25278265
- [Derived] Zhang J, Wang X, Wang X, Hui A, Wu Z, Tian L, Xu C, Yang Y, Zhang W, Hu X. Phase 1a study of the CDK4/6 inhibitor, FCN-437c, in Chinese patients with HR + /HER2- advanced breast cancer. Invest New Drugs. 2021 Dec;39(6):1549-1558. doi: 10.1007/s10637-021-01133-2. Epub 2021 Jun 9. PMID 34109484
- Available data/document: ICH topic S9 - nonclinical evaluation for anticancer pharmaceuticals. 2009: ICH topic S9 — https://database.ich.org/sites/default/files/S9_Guideline.pdf
- Available data/document: label for IBRANCE® (palbociclib) capsules: IBRANCE® (palbociclib) capsule — https://www.accessdata.fda.gov/drugsatfda_docs/label/2015/207103s000lbl.pdf
- Available data/document: label for IBRANCE® (palbociclib) tablets,: IBRANCE® (palbociclib) tablets — https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/212436lbl.pdf
- Available data/document: Label for KISQALI® (ribociclib) tablets: KISQALI® (ribociclib) tablets — https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/209092s005lbl.pdf
- Available data/document: ICH Topic E6 (R1) Guideline for Good Clinical Practice: ICH Topic E6 (R1) — https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e6-r1-guideline-good-clinical-practice_en.pdf
- Available data/document: ICH Topic E9 Statistical Principles for Clinical Trials: ICH Topic E9 — https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e-9-statistical-principles-clinical-trials-step-5_en.pdf